CLINICAL TRIAL: NCT05452902
Title: The Effects of Exercise and Nutrition Interventions on Platinum Chemotherapy-induced Peripheral Neuropathy and Interoceptive Brain Circuitry (R21)
Brief Title: Exercise and Nutrition Interventions for Platinum Chemotherapy-induced Neuropathy R21
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Out of time and study resources
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ian Kleckner, PhD, MPH, Associate Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HP-00100000; R21CA259422 (NIH)
Record Dates: First submitted 2022-07-06; First posted 2022-07-11 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy
Keywords: Chemotherapy; Brain; Exercise; Nutrition
MeSH Terms: conditions — Motor Activity | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXCAP Exercise (Experimental): Exercise for Cancer Patients (EXCAP©®) involves face-to-face instruction and a prescription for an at-home progressive walking and resistance exercise program.
  Interventions: Behavioral: EXCAP Exercise
- Nutrition Education (Active Comparator): Nutrition education involves equal time and attention as the exercise arm, but the content covers nutrition for cancer patients and lacks an exercise prescription.
  Interventions: Behavioral: Nutrition Education

INTERVENTIONS:
Behavioral: EXCAP Exercise — 12 weeks of at-home walking and resistance exercise.
  Arms: EXCAP Exercise
Behavioral: Nutrition Education — 12 weeks of implementing eating tips and tracking food.
  Arms: Nutrition Education

SUMMARY:
Chemotherapy-induced peripheral neuropathy (CIPN) is a highly prevalent and severe side-effect of platinum-based chemotherapy, often used to treat gastrointestinal cancers. Unfortunately there are very limited treatments for CIPN. This is a phase II randomized controlled trial to test the preliminary efficacy of exercise vs. nutrition education on CIPN, to systematically investigate the potential roles of inflammation and interoception, and to obtain data with a more accurate effect size to inform a future study.

ELIGIBILITY:
Inclusion criteria (subjects must…)

1. Have a diagnosis of cancer
2. Be scheduled to receive platinum chemotherapy (specifically oxaliplatin or cisplatin) without other neurotoxic chemotherapy (taxanes, bortezomib, thalidomide). Patients may be enrolled before their first (preferred), second, or third infusion of neurotoxic chemotherapy
3. Be able to read English
4. Be ≥18 years

Exclusion criteria (subjects must not…)

1. Be performing regular exercise, which is any planned physical activity (e.g., brisk walking, aerobics, jogging, bicycling, swimming, rowing, weight lifting, resistance training, yoga, pilates, etc.) performed to increase physical fitness. To be considered exercise, physical activity should be performed 3-5 times per week for 20-60 minutes per session and should be done at a level that increases your breathing rate and causes you to break a sweat.
2. Have physical limitations (e.g., cardiorespiratory, orthopedic, central nervous system) that contraindicate participation in maximal physiological fitness testing and a low/moderate intensity home-based walking and progressive resistance exercise program.
3. Have planned surgery or radiation treatment in the 12 weeks after baseline.

Additional exclusion criteria only for patients completing MRI (approximately 40 of 60 enrolled subjects; subjects must not…)

1. Have current or prior cancer in the spine, brainstem, or brain (to allow standard brain MRI analysis)
2. Have contraindications for MRI scanning (pacemaker, ferrous metal implants, pregnancy, etc. note that most port-a-caths are safe for MRI scanning)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-01-19 (Actual); Primary Completion 2025-09-25 (Actual); Study Completion 2025-09-25 (Actual)

PRIMARY OUTCOMES:
CIPN-20 sensory subscale | Time point 2 (approximately 6 weeks), controlling for baseline value
  CIPN-20 sensory subscale (Postma et al 2005). The subscale includes 9 questions, each rated 1-4, and the score ranges from 9-36 with larger values reflecting more severe (worse) symptoms of chemotherapy-induced peripheral neuropathy (CIPN).

SECONDARY OUTCOMES:
CIPN-20 sensory subscale | Time point 2 (approx. 6 weeks) or time point 3 (approx. 12 weeks) or time point 4 (approx. 24 weeks), controlling for baseline
  CIPN-20 sensory subscale (Postma et al 2005). The subscale includes 9 questions, each rated 1-4, and the score ranges from 9-36 with larger values reflecting more severe (worse) symptoms of chemotherapy-induced peripheral neuropathy (CIPN).
Sensory, motor, and autonomic symptoms of CIPN | Time point 2 (approx. 6 weeks) or time point 3 (approx. 12 weeks) or time point 4 (approx. 24 weeks), controlling for baseline
  CIPN-20 total score (Postma et al 2005). The score includes 20 questions, each rated 1-4, and the score ranges from 20-80 with larger values reflecting more severe (worse) symptoms of chemotherapy-induced peripheral neuropathy (CIPN).
Sensory loss | Time point 2 (approx. 6 weeks) or time point 3 (approx. 12 weeks), controlling for baseline
  Finger and toe tactile sensitivity using monofilaments
Cold-induced pain | Time point 2 (approx. 6 weeks) or time point 3 (approx. 12 weeks), controlling for baseline
  Finger cold sensitivity using thermode
Numbness and tingling | Time point 2 (approx. 6 weeks) or time point 3 (approx. 12 weeks), controlling for baseline
  Patient-reported severity of numbness/tingling (0-10). A larger value reflects more severe (worse) symptoms of chemotherapy-induced peripheral neuropathy (CIPN).

OTHER OUTCOMES:
Neuropsychological function | Time point 2 (approx. 6 weeks) or time point 3 (approx. 12 weeks), controlling for baseline
  Brain connectivity via functional magnetic resonance imaging
Immunological function | Time point 2 (approx. 6 weeks) or time point 3 (approx. 12 weeks), controlling for baseline
  Inflammatory cytokine concentration via ELISA (IL-6, IL-10, etc.)
Musculoskeletal function | Time point 2 (approx. 6 weeks) or time point 3 (approx. 12 weeks), controlling for baseline
  Strength via handgrip dynamometer test
Cardiovascular function | Time point 2 (approx. 6 weeks) or time point 3 (approx. 12 weeks), controlling for baseline
  Distance walked in six-minute walk test

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland Medical System, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
* First, we will conduct our primary analyses (Aims 1-4) on the data collected and publish our results with a group of researchers determined by the PI: Dr. Kleckner. Our team has already worked together to develop our study design, analysis plan, dissemination plan, etc. and we want to be the ones to publish our findings.
  * Second, after the primary analyses (Aims 1-4) have been published (or at the discretion of the PI), we welcome collaboration with others who want to analyze our data as long as we are offered an opportunity for co-authorship and collaboration (not simply passing the data off to another research group). We may or may not accept the invitation for co-authorship depending on the timing and nature of the research.
  * Third, if there are questions about the validity of our published findings and other research groups want to perform an independent analysis that they feel would be compromised by our co-authorship or collaboration, then we are open to that possibility.
Time Frame: See above plan
Access Criteria: Researchers analyzing our data must adhere to the following agreement (or similar), which will be presented in writing and signed and dated:
  * They will not transfer the data to another party (i.e., all data requests come to the study PI, Dr. Kleckner)
  * They will maintain the security and privacy of the data (secure data servers, password-protected computers, secure data transfer methods, etc.).
  * They will acknowledge our funding sources that supported collection of the data (including this R21)
  * They will offer collaboration and co-authorship unless that would be deemed inappropriate for ethical reasons (e.g., conducting an independent analysis)
  * They will notify the study PI, Dr. Kleckner of dissemination (abstracts, manuscripts, etc.)
  * They will provide regular updates to Dr. Kleckner on progress analyzing the data

REFERENCES:
- [Background] Postma TJ, Aaronson NK, Heimans JJ, Muller MJ, Hildebrand JG, Delattre JY, Hoang-Xuan K, Lanteri-Minet M, Grant R, Huddart R, Moynihan C, Maher J, Lucey R; EORTC Quality of Life Group. The development of an EORTC quality of life questionnaire to assess chemotherapy-induced peripheral neuropathy: the QLQ-CIPN20. Eur J Cancer. 2005 May;41(8):1135-9. doi: 10.1016/j.ejca.2005.02.012. Epub 2005 Apr 14. PMID 15911236